CLINICAL TRIAL: NCT04952636
Title: A Prospective Comparative Study of Arthroscopic and Open Surgery in Chinese Unique Inlay Bristow Procedure
Brief Title: A Prospective Comparative Study of Arthroscopic and Open Surgery in Cuistow Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2020294
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-07

CONDITIONS: Shoulder Dislocation
Keywords: recurrent anterior shoulder dislocation; Bristow-Latarjet procedure; arthroscopy
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic Cuistow (Experimental): Patients who receive arthroscopic Cuistow procedure
  Interventions: Procedure: arthroscopic Cuistow
- Open Cuistow (Experimental): Patients who receive open Cuistow procedure
  Interventions: Procedure: open Cuistow

INTERVENTIONS:
Procedure: arthroscopic Cuistow — peforming the Cuistow Procedure under arthroscopy
  Arms: Arthroscopic Cuistow
Procedure: open Cuistow — peforming the Cuistow Procedure with the traditional open process
  Arms: Open Cuistow

SUMMARY:
To evaluate the clinical outcomes of arthroscopic and open Chinese Unique Inlay Bristow procedure in treating recurrent anterior shoulder instability.

DETAILED DESCRIPTION:
Recurrent anterior dislocation of the shoulder joint is a common disorder of the shoulder joint. Patients with recurrent anterior dislocation of the shoulder severely affect movement and quality of life, and severe cases can lead to severe dysfunction of the shoulder joint. Nowadays, arthroscopic Bankart surgery is routinely used to treat such patients. However, the recurrence rate of shoulder dislocation with conventional arthroscopic Bankart repair is high in professional athletes with very high levels of athleticism and in complex patients with large glenoid bone defects. For this population, coracoid transfer surgery (Bristow-Latarjet procedure) is currently considered to have better efficacy.

The Latarjet procedure is now relatively well established internationally; however, this technique has a large osteotomy block and uses two hollow screws to fix the bone block. This is very traumatic and cannot be used in patients with small coracoid, and there is a high incidence of postoperative bone resorption of the bone block, and in the event of severe bone resorption, the screws left behind are more damaging to the subscapularis tendon. In contrast, the Bristow procedure is relatively less invasive, but the early healing rate of the grafted bone block is lower than that of the Latarjet procedure. In response to this problem, the group improved the Bristow procedure in a previous clinical study by using an embedded technique to fix the bone block, which is the first of its kind in the world, and the investigators named it the Chinese Unique Inlay Bristow (Cuistow) procedure. The description and clinical results of this procedure have been accepted by the American Journal of Sports Medicine, and the technique is now a routine procedure in our department.

There is still some debate as to whether the classical coracoid procedure should be performed arthroscopically or open. Open surgery is more traumatic, but relatively easy to perform, with a shorter operative time and a shorter learning curve to master the technique; arthroscopic surgery is less traumatic, with faster recovery, but relatively more expensive and requires higher surgical skills. Some studies have concluded that there is no significant difference between the two in terms of long-term postoperative outcomes and complications. In our previous study, the investigators found that the use of our first " Mortise and Tenon structure " bone displacement fixation resulted in better early postoperative stability and higher postoperative bone healing rates than the traditional coracoid transfer procedure. However, it is unknown whether there is a difference in clinical outcomes and postoperative bone healing rates using open surgery compared to arthroscopic surgery.

In this study, a prospective observational study was conducted in which the advantages and disadvantages of arthroscopic and open surgery for Cuistow procedure were explained to the patient before surgery, and then the patient chose one of the surgical approaches according to his or her own wishes. The functional recovery and bone resorption of the two groups were compared, and the two surgical approaches were evaluated to determine whether there were significant differences in postoperative bone healing rates and clinical outcomes between the two surgical approaches.

In conclusion, the aim of this study was to evaluate the advantages and disadvantages of the two surgical approaches through a comparative study. The investigators wish to provide a complete systematic solution for the treatment of difficult and complex recurrent anterior shoulder dislocations, and to provide an effective remedy for cases of recurrence after Bankart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. a glenoid defect ≥10%
2. contact sport athletes with a glenoid defect < 10%
3. failure after Bankart repair.

Exclusion Criteria:

1. epilepsy
2. multidirectional shoulder instability
3. concomitant other lesions including rotator cuff tear, symptomatic acromioclavicular joint pathology or pathological involvement of the long head of the biceps

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
ASES score | 2 years after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is the most commonly used score to describe the function of patients' shoulder joints, ranging from 0 to 100. The higher the score, the better the function of patients' shoulder joints.
pain VAS score | 2 years after surgery
  The visual analog scale (VAS) for pain score is the most commonly used to describe pain levels in patients, ranging from 0 to 10, with a higher score indicating more intense pain.

SECONDARY OUTCOMES:
Active shoulder ranges of motion | 2 years after surgery
  internal rotation at the side, and external and internal rotation at 90° of abduction
Bone block position | immediately after surgery
  Bone block position was evaluated using postoperative CT scans.The ideal position of the bone block was defined as flush to the anterior glenoid rim in the axial view and 4 o'clock in the En face view. The bone block was considered too lateral if it went beyond the glenoid rim by more than 5 mm and it was judged to be too medial if it was medial to the rim by more than 5 mm.
Bone union | 3 months after surgery
  Graft union with the glenoid was assessed using postoperative CT scans. ''Bony union'' of the transplant was defined as no radiolucent zone; ''fibrous union,'' when the transplant had a radiolucent zone of less than 5 mm; and ''migration,'' when the zone
Bone union | 2 years after surgery
  Graft union with the glenoid was assessed using postoperative CT scans. ''Bony union'' of the transplant was defined as no radiolucent zone; ''fibrous union,'' when the transplant had a radiolucent zone of less than 5 mm; and ''migration,'' when the zone

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, Study Chair — Peking University Third Hospital
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No